CLINICAL TRIAL: NCT01571219
Title: An Open-Label, Single-Arm, Extension Study to Demonstrate Long-Term Efficacy and Safety of CT-P13 When Co-Administered With Methotrexate in Patient With Rheumatoid Arthritis Who Were Treated With Infliximab(Remicade or CP-P13) in Study CT-P13 3.1
Brief Title: An Extension Study to Demonstrate Long-Term Efficacy and Safety of CT-P13 When Co-administered With Methotrexate in Patient With Rheumatoid Arthritis Who Were Treated With Infliximab (Remicade or CT-P13) in Study CT-P13 3.1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celltrion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT-P13 3.2; 2011-004468-31 (EudraCT Number)
Record Dates: First submitted 2012-03-23; First posted 2012-04-05 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Rheumatoid Arthritis
Keywords: RA; Biosimilar
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CT-P13 (Experimental)
  Interventions: Biological: Infliximab

INTERVENTIONS:
Biological: Infliximab — CT-P13(3mg/kg) administered as a 2-hour IV infusion per dose co-administered with methotrexate between 12.5 to 25 mg/week, oral or parenteral dose (dose and route must be maintained from Study CT-P13 3.1 and be maintained from the beginning to the end of the extension study) and folic acid(≥5mg/week, oral dose)

SUMMARY:
CT-P13 (Infliximab) is a monoclonal antibody currently being developed by CELLTRION, Inc. This open-label, single-arm, multicenter, multiple single dose intravenous (IV) infusion, efficacy, and safety extension study of the Phase 3 Study CT-P13 3.1 is designed to assess the long-term efficacy and safety of multiple doses of CT-P13.

ELIGIBILITY:
Inclusion Criteria:

* Patient who has completed the scheduled visits, including the End-of-Study Visit, in Study CT-P13 3.1
* Patient who has not had any major protocol violation in Study CT-P13 3.1
* Patient is permitted to enter the extension study if, in the option of their general practitioner or the investigator, the patient will continue to gain benefit from treatment in the extension study. Local guidelines for patient treatment will be followed

Exclusion Criteria:

* Patient who has been withdrawn from Study CT-P13 3.1 for any reason
* Patient who, at the time of providing informed consent, has any ongoing medical issues such as serious adverse events (SAEs) or intolerance issues that mean continuation in this extension study could be detrimental to their health, in the opinion of the investigator
* Patient who plans to participate in a study with an investigational drug during the period of this extension study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2012-03; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Long term efficacy evaluated by American College of Rheumatology(ACR) criteria and Long term safety evaluated by immunogenicity and clinical laboratory test | Up to week 40

CONTACTS AND LOCATIONS:
Overall Officials: Dae Hyun Yoo, M.D., Ph.D., Study Director — Hanyang University
Locations (1):
- Hanyang University Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Yoo DH, Prodanovic N, Jaworski J, Miranda P, Ramiterre E, Lanzon A, Baranauskaite A, Wiland P, Abud-Mendoza C, Oparanov B, Smiyan S, Kim H, Lee SJ, Kim S, Park W. Efficacy and safety of CT-P13 (biosimilar infliximab) in patients with rheumatoid arthritis: comparison between switching from reference infliximab to CT-P13 and continuing CT-P13 in the PLANETRA extension study. Ann Rheum Dis. 2017 Feb;76(2):355-363. doi: 10.1136/annrheumdis-2015-208786. Epub 2016 Apr 29. PMID 27130908